CLINICAL TRIAL: NCT02070809
Title: Multicenter Clinical Randomized Controlled Trials on Rapid Construction of Tissue-engineered Skin for Repairing Wounds
Brief Title: Rapid Construction of Tissue-engineered Skin for Repairing Wounds
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Zhu Jiayuan, Professor, vice director of surgery, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013001
Record Dates: First submitted 2014-02-22; First posted 2014-02-25 (Estimated); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Wound
Keywords: wound; tissue-engineered skin
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tissue-engineered skin method (Experimental): This method is composite of skin grafting over human acellular dermal matrix scaffold the investigators used before with skin basal cell as seed cells, moreover it was finished in the surgery without culturing the cells
  Interventions: Procedure: tissue-engineered skin method
- split-thickness skin graft method (Active Comparator): This method is traditional split-thickness skin graft
  Interventions: Procedure: split-thickness skin graft method

INTERVENTIONS:
Procedure: tissue-engineered skin method — This method is composite of skin grafting over human acellular dermal matrix scaffold the investigators used before with skin basal cell as seed cells, moreover it was finished in the surgery without culturing the cells
  Arms: tissue-engineered skin method
Procedure: split-thickness skin graft method — This method is traditional split-thickness skin graft
  Arms: split-thickness skin graft method

SUMMARY:
A wound comprises a break in epithelial continuity and disruption of structure and function of underlying tissues, the treating and repairing is always a great challenge in clinical practice. The complex healing process make the wound easy to get a tendency of nonhealing and result in a heavy burden of life quality. Nowadays surgical repairing is still the main method, but there was still no effective and satisfy outcomes. Because none of the treatments could repair skin both on structure and function. Now the investigators provide a quick and effective method to rebuilt complete structure and function of the skin based on tissue-engineered skin technology. To further test the efficacy and safety of this new method, the investigators propose a prospective randomized controlled multicenter trial to compare this method with traditional skin graft.

DETAILED DESCRIPTION:
A wound comprises a break in epithelial continuity and disruption of structure and function of underlying tissues, the treating and repairing is always a great challenge in clinical practice. The complex healing process make the wound easy to get a tendency of nonhealing and result in a heavy burden of life quality. Nowadays surgical repairing is still the main method, such as traditional split-thickness skin graft, flap transplantation or tissue-engineered substitute transplantation. However, none of these methods could have effective and satisfy outcomes. Because none of these treatments could repair skin on both structure and function. Therefore, as a new treating technology the tissue-engineered skin has been widely used recently and shows good response. As a consequence, the investigators provide a quick and effective method to rebuilt complete structure and function of the skin based on tissue-engineered skin technology. This method is composite of skin grafting over human acellular dermal matrix scaffold the investigators used before with skin basal cell as seed cells, moreover it was finished in the surgery without culturing the cells and could greatly reduce the time. To further test the efficacy and safety of this new method, the investigators propose a prospective randomized controlled multicenter trial to compare this method with traditional skin graft. If this method could actually increase wound take rate, improve the skin quality and restore skin function in some extent, it should resolve the problem of wound repair to a large extent.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who need to skin graft to repair the wound
* Subjects signed the informed consent in the day of the age of not more than 81 years old (for minors, legal guardian should be signed)
* Stable vital signs, regular examination showed that subjects could tolerate surgery
* Subjects' mental state are good, could follow the doctor's advice, visit on a regular basis
* Understanding and willing to participate in this clinical trial and signed informed consent
* All women subjects must agree to take effective contraceptive measures in the six months study period, and without pregnancy before participate in the treatment
* No other serious diseases conflicts with the trail
* Wound size between 3 cm2 and 100 cm2, no limited to location

Exclusion Criteria:

* Allergic constitution of enzyme
* Severe uncontrolled disease or acute systemic infections and complication with other serious heart, lung disease, encephalopathy and other organs or have a rapid progress or terminal disease
* Subjects with mental illness
* Subjects could not cooperate with the clinical trial personnel to finish trials
* Existing disease (malignant tumor, autoimmune disease) or require the use of drugs (high-dose glucocorticoids, which is defined as accepting 40 mg or more daily prednisone or prednisone amount, period of two weeks or more) will affect the healing of the wound
* For HIV positive patients, clinical diagnosis of patients with AIDS or the screening phase of neutrophil count (ANC) absolutely < 1000 cells/mm3
* Subjects could not tolerate surgery
* Subjects are unlikely to survive in the study period
* The investigators think that who should not be included
* Subjects are in or participated in other clinical researchers over the past 12 weeks
* Subjects are participated in this trial at any time in the past

Max Age: 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 386 (Estimated)
Dates: Start 2013-12 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
healing rate | postsurgery week 4
  the percentage of subjects that achieved complete wound closure, complete wound closure is defined as skin complete reepithelialization without drainage or dressing requirements.

SECONDARY OUTCOMES:
wound reducing rate | postsurgery week 4
  the rate of wound reducing based on week 4 after surgery

OTHER OUTCOMES:
recurrence rate | postsurgery month 6
  the incidence of ulcer recurrence at postsurgery month 6

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Zhu, doctor, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China